CLINICAL TRIAL: NCT00855842
Title: Pilot Study of the Addition of Osmotic Dilators to Preparation Prior to Labor Induction Abortion
Acronym: DAIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate enrollment
Sponsor: Boston University (Other)
Responsible Party: Lynn Borgatta MD, Boston University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIS
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-06

CONDITIONS: Abortion, Induced
Keywords: second trimester abortion; labor induction abortion; second trimester medical abortion; pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- osmotic dilator (Experimental): osmotic dilator
  Interventions: Device: osmotic dilator insertion

INTERVENTIONS:
Device: osmotic dilator insertion — osmotic dilators are placed in the cervix to cause cervical dilation
  Other Names: laminaria; Dilapan

SUMMARY:
One the day prior to medical abortion (labor induction) in the second trimester, insertion of osmotic dilators is added to the routine procedures. The study is to see whether the addition of dilators decreases the abortion time (time for the pregnancy to be expelled)

DETAILED DESCRIPTION:
This is a pilot study and is an uncontrolled, non-randomized series. Women having a medical abortion in second trimester undergo several procedures the day before the medication to cause contractions occurs. On the day before admission, they take mifepristone orally, and have a feticidal injection. to this would be added the insertion of cervical osmotic dilators (the intervention). On the day of induction, the dilators would be removed and misoprostol started to cause contractions. We are hoping the median abortion time will drop from the present 9-10 hours to 4-6 hours. women who do not abort in 6 hours will have option of surgical completion of the abortion (dilation and evacuation) if medically appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Requesting abortion 19-23 weeks
* No contraindication to induction abortion

Exclusion Criteria:

* Fetal demise
* Ruptured membranes
* Evidence of pelvic infection
* Inability to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Borgatta, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women requesting abortion at 19-23 weeks were eligible to enroll if they were able to consent and had no contraindications to medical abortion. Women were informed of the study after all counseling for abortion was completed and after they had given consent for abortion
Pre-assignment Details: Women were eligible for study intervention if they had singleton pregnancy with intact membranes, without signs of infection.
Period: Overall Study
Arm/Group | Osmotic Dilator
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Osmotic Dilator
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Length of Medical Abortion
Description: This is the time elapsed from the first dose of misoprostol (the agent to induce abortion) and expulsion of the fetus
Time Frame: hours since the start of medical abortion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Osmotic Dilator
Number analyzed (Participants) | 4
hours | 7 (5)

ADVERSE EVENTS:
Arm/Group | Osmotic Dilator
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The study was terminated early because the clinical facility changed and eligible patients were not seen at the facility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No